CLINICAL TRIAL: NCT06504654
Title: Interoception and Eating Behaviors in Children
Acronym: I-EAT
Status: Recruiting | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Emily Hohman, Associate Research Professor, Penn State University
Other Study IDs: STUDY00024712
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity, Childhood; Eating Behavior
Keywords: interoception; eating behavior; ghrelin
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva samples will be collected at fasting and 30, 60, and 90 minutes after a meal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to examine how individual differences in interoception (the ability to sense, interpret, and act on bodily feelings like hunger, fullness, thirst, hot, cold, etc.) relate to eating behaviors in children ages 7-10 years. Findings will inform whether interventions targeting interoceptive awareness may be helpful for prevention of obesity and related chronic diseases.

DETAILED DESCRIPTION:
The overall goal of this project is to examine if interoception (the process by which internal bodily states, like hunger and fullness, are sensed, integrated, interpreted, and regulated) is associated with BMI and obesity-related eating behaviors in children age 7-10 years. The specific aims are:

Aim 1: Determine associations between interoception and non-homeostatic eating H1: Multi-systems measures of interoceptive awareness (e.g., heartbeat perception, gastric interoception, self-reported interoceptive awareness) will be inversely associated with intake (kcal) in the eating in the absence of hunger (EAH) task

Aim 2: Assess salivary ghrelin and leptin as interoceptive signals of hunger/satiety H1: Children with greater postprandial suppression of ghrelin will eat less in the EAH task H2: Children with greater postprandial suppression of ghrelin will have better interoceptive awareness H3: Children with higher leptin will exhibit less sensitivity to changes in ghrelin

Aim 3 (Exploratory): Identify interoceptive phenotypes that may predict obesity risk Using k-means cluster analysis, we aim to identify subgroups of individuals who exhibit different combinations of interoceptive variables. We will then examine differences in eating behavior and weight between clusters.

Participants will attend two study visits at the Clinical Research Center at Penn State University Park campus. At the first visit, children will have their height, weight, and body composition measured, complete measures of interoception, and complete surveys/interview. Parents will complete a survey. At the second visit, children will eat a meal, taste snacks, provide saliva samples, and play cognitive games on a tablet.

ELIGIBILITY:
Inclusion Criteria:

* Child must be 7-10 years of age
* Participating parent must be at least 18 years of age, but there is no upper age limit
* Able to understand and answer questions in English

Exclusion Criteria (all applicable to child only):

* BMI for age <5th percentile
* Monogenic obesity condition (e.g., Prader Willi syndrome)
* Autism/autism spectrum disorder
* Developmental delay
* Eating disorder
* Diabetes
* Heart condition
* Taking medications impacting appetite (e.g., stimulants, weight control medications)
* Any other condition significantly impacting growth, eating behavior, or cardiac function
* Allergy or dietary restriction to study foods
* Severe/untreated oral/dental health problems
* Orthodontic procedure or adjustment of braces within the past omonth
* Oral surgery or major oral/dental procedure within past month
* Had an x-ray within the past month

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children 7-10 years old and their parents
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Kcal consumed in the Eating in the Absence of Hunger protocol | Visit 2 (1-3 weeks after enrollment at Visit 1)
  Children will be provide with an array of snacks following a meal and will have 10 minutes to consume any snacks that they would like. Intake will be measured by pre- and post-weighing snacks

SECONDARY OUTCOMES:
Pattern of salivary ghrelin in response to a meal | Visit 2 (1-3 weeks after enrollment at Visit 1)
  Children will provide saliva samples at fasting, +30 minutes, +60 minutes, and +90 minutes from start of a meal, which will be analyzed for active ghrelin
Pattern of salivary leptin in response to a meal | Visit 2 (1-3 weeks after enrollment at Visit 1)
  Children will provide saliva samples at fasting, +30 minutes, +60 minutes, and +90 minutes from the start of a meal, which will be analyzed for leptin
Heart beat counting accuracy | Visit 1 (Enrollment)
  Participants will be fitted with a heart rate monitor and will be asked to count their heartbeat over several time intervals. Reported counts will be compared to measured heart rate to determine percent accuracy
Gastric interoception | Visit 1 (Enrollment)
  Children will be asked to drink plain water until their stomach feels 'just right', and then will be asked to drink further water until their stomach feels maximally full. The amount of water consumed in each phase will be measured by changes in weight of the water bottle. The ratio of the two volumes is a measure of gastric interoception that is not confounded by stomach capacity
Multidimensional Assessment of Interoceptive Awareness (MAIA)-youth version | Visit 1 (Enrollment)
  Children will complete a questionnaire via interview to assess their perception of their interoceptive awareness

CONTACTS AND LOCATIONS:
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared in a repository at the end of the study
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be shared at the conclusion of the funding period (July 2026)
Access Criteria: Data will be shared in accordance with access criteria of the selected repository (to be determined)